CLINICAL TRIAL: NCT02365220
Title: Smartphone Application, Mood and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: University of Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UNIBAS-MMH-SMA1
Record Dates: First submitted 2015-02-03; First posted 2015-02-18 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Smartphone Application; Placebo Effect; Mood; Stress
MeSH Terms: interventions — Longitudinal Studies

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- No expectancy (control) (Active Comparator): No expectancy instruction with regard to the efficacy of the daily smartphone-based training
  Interventions: Behavioral: No expectancy (control)
- Prospective expectancy (Experimental): Prospective expectancy instruction ("Training will have an effect on...") with regard to the efficacy of the daily smartphone-based training
  Interventions: Behavioral: Prospective expectancy
- Retrospective expectancy (Experimental): Retrospective expectancy instruction ("Training already had an effect on...") with regard to the efficacy of the daily smartphone-based training
  Interventions: Behavioral: Retrospective expectancy
- Prospective and retrospective expectancy (Experimental): Prospective ("Training will have an effect on...") and retrospective ("Training already had an effect on...") expectancy instruction with regard to the efficacy of the daily smartphone-based training
  Interventions: Behavioral: Prospective and retrospective expectancy

INTERVENTIONS:
Behavioral: No expectancy (control) — No expectancy instruction with regard to the efficacy of the daily smartphone-based training (exposition to either mock sound or color)
  Arms: No expectancy (control)
Behavioral: Prospective expectancy — Prospective expectancy instruction ("Training will have an effect on...") with regard to the efficacy of the daily smartphone-based training (exposition to either mock sound or color)
  Arms: Prospective expectancy
Behavioral: Retrospective expectancy — Retrospective expectancy instruction ("Training already had an effect on...") with regard to the efficacy of the daily smartphone-based training (exposition to either mock sound or color)
  Arms: Retrospective expectancy
Behavioral: Prospective and retrospective expectancy — Prospective ("Training will have an effect on...") and retrospective ("Training already had an effect on...") expectancy instruction with regard to the efficacy of the daily smartphone-based training (exposition to either mock sound or color)
  Arms: Prospective and retrospective expectancy

SUMMARY:
The purpose of this study is to investigate the placebo effect in a smartphone-based training, ostensibly designed to improve mood and perceived stress by daily exposition to either mock sound or color.

DETAILED DESCRIPTION:
The overall goal of the outlined study is to investigate the placebo effect in a smartphone-based training, ostensibly designed to improve mood and perceived stress by daily exposition to either mock sound or color. During 14 days, subjects will participate in regular daily training sessions. During another 6 days, subjects will transfer the smartphone-based training to daily life.

ELIGIBILITY:
Inclusion Criteria:

* Access to smartphone during study period

Exclusion Criteria:

* Severe visual impairment
* Dyschromatopsia
* Severe defective hearing
* Regular intake of medication (excl. contraceptives)
* Severe mental disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-02; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Change in mood (Assessed via Multidimensional Mood State Questionnaire) | Pre- and post-training, during 20 days of training
  Assessed via Multidimensional Mood State Questionnaire
Change in perceived stress | Pre- and post-training, during 20 days of training
  Assessed via State-Trait-Anxiety Inventory; Visual Analog Scale

SECONDARY OUTCOMES:
Emotional state (Assessed via Self-Assessment-Manikin scales) | Post-training, during 20 days of training
  Assessed via Self-Assessment-Manikin scales after exposition to affective pictures taken from International Affective Picture System

OTHER OUTCOMES:
Efficacy expectancy (Assessed via Credibility Expectancy Questionnaire) | Post-training, training day 1, 7, 14, 20
  Assessed via Credibility Expectancy Questionnaire
Feedback on adverse events during the daily training session (Number of subjects reporting an adverse event) | Post-training, last training day (day 20)
  Number of subjects reporting an adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Gunther Meinlschmidt, Prof. Dr., Principal Investigator — University of Basel, Department of Psychology, Division of Clinical Psychology and Epidemiology
Locations (1):
- University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Stalujanis E, Neufeld J, Glaus Stalder M, Belardi A, Tegethoff M, Meinlschmidt G. Induction of Efficacy Expectancies in an Ambulatory Smartphone-Based Digital Placebo Mental Health Intervention: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 17;9(2):e20329. doi: 10.2196/20329. PMID 33594991